CLINICAL TRIAL: NCT03691155
Title: The Feasibility of Following the Crohn's Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: LRS-17/18-7313
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases; Dietary Modification
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The Crohn's Diet — All recruited participants will be educated on the Crohn's Diet and instructed to adhere to the study diet for 14 days.

SUMMARY:
A research team from King's College London are investigating how diet can be used as a treatment for Crohn's disease. The investigators have designed a new diet and eventually wish to test whether the diet can be used to manage Crohn's disease and reduce gut inflammation. Before doing this, the investigators need to find out how practical it is for people to follow the diet for 14 days by conducting this 'feasibility' study. A feasibility study is a small study that aims to highlight any issues before informing the design of a larger research trial.

The diet the investigators have designed is called the Crohn's Diet. The evidence for this diet is based on recent research which suggests that certain food ingredients may be involved in triggering gut inflammation.

The study's primary aim is to assess the practicalities of following the Crohn's Diet. It will also assess compliance to the Crohn's Diet and if following it changes the nutritional balance from the normal diet.

ELIGIBILITY:
Inclusion Criteria will include:

1. Adults aged ≥18 years with a diagnosis of Crohn's disease
2. Stable Crohn's disease (as defined as self-reported: no change in Crohn's disease medication in the last 3 months; no Crohn's disease surgery in the last 6 months; no hospital admissions related to Crohn's disease in the last 6 months; no new perianal Crohn's disease in the last 6 months).
3. Individuals with a Body Mass Index (BMI) of ≥ 18.5 kg/m2
4. Individuals able to give informed consent
5. Individuals able to understand and read English
6. Individuals willing to provide consent in this study which involves a dietary change for 14 days

Exclusion Criteria will include:

1. Unexplained/unintentional weight loss in the past 6 months
2. Major co-morbidities; for example, diabetes, coeliac disease, major active psychiatric conditions or current eating disorders.
3. Current Crohn's disease therapy with any of the following: corticosteroids, exclusive or partial enteral nutrition (liquid nutrition), and any participants prescribed oral nutrition supplements for nutrition support.
4. Individuals who report to be pregnant or lactating
5. Individuals with specific, complex dietary needs (based on the dietitian's judgment), such as multiple food allergies, in which the additional burden of the Crohn's Diet would pose a nutrition risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of following the Crohn's Diet: questionnaire | Throughout the 14-day intervention
  Method: Collation of participant feedback during the Crohn's Diet and administer diet feasibility questionnaire. This questionnaire uses an adapted Education Method Usability Scale (Bangor et al. 2008) ('strongly agree' to 'strongly disagree' style scale) and open questions.

SECONDARY OUTCOMES:
Acceptability of following the Crohn's Diet: questionnaire | Throughout the 14-day intervention and within one week of completing the intervention
  Method: Administer questionnaires on diet acceptability, including the Food-Related Quality of Life in Inflammatory Bowel Disease questionnaire (Hughes et al 2016).
Participant compliance to the Crohn's Diet | Throughout the 14-day intervention
  Method: Dietitian monitoring of compliance during the trial. A 7-day food diary will quantify compliance alongside a questionnaire which explores reasons for potential non-compliance.
Impact of the Crohn's Diet on habitual dietary intake | One week before the intervention and throughout the 14-day intervention
  Method: 7-day food diaries to compare nutrient intake and explore changes in dietary patterns.
Impact of the Crohn's Diet on BMI | One week before the intervention and within one week of completing the 14-day intervention
  Method: Participants will undergo anthropometric assessment, including weight and height to report BMI.
Impact of the Crohn's Diet on gastrointestinal symptoms | One week before the intervention and within one week of completing the 14-day intervention
  Method: Administer the PRO-2 questionnaire (Khanna et al 2015).
Impact of the Crohn's Diet on perceived disease control | One week before the intervention and within one week of completing the 14-day intervention
  Method: Administer questionnaires, including the Inflammatory Bowel Disease Control-8 questionnaire (IBD-C-8) (Bodger et al. 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Whelan, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No